CLINICAL TRIAL: NCT04034927
Title: A Phase II Randomized Trial of Olaparib Versus Olaparib Plus Tremelimumab in Platinum-Sensitive Recurrent Ovarian Cancer
Brief Title: Testing the Addition of an Immunotherapy Drug, Tremelimumab, to the PARP Inhibition Drug, Olaparib, for Recurrent Ovarian, Fallopian Tube or Peritoneal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-04829; NCI-2019-04829 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY021 (Other: NRG Oncology); NRG-GY021 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Results first posted 2023-10-13 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Fallopian Tube Endometrioid Tumor; Fallopian Tube High Grade Serous Adenocarcinoma; Malignant Ovarian Endometrioid Tumor; Ovarian High Grade Serous Adenocarcinoma; Platinum-Sensitive Fallopian Tube Carcinoma; Platinum-Sensitive Ovarian Carcinoma; Platinum-Sensitive Primary Peritoneal Carcinoma; Primary Peritoneal High Grade Serous Adenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Fallopian Tube Endometrioid Adenocarcinoma; Recurrent Ovarian Endometrioid Adenocarcinoma; Recurrent Ovarian Serous Adenocarcinoma; Recurrent Primary Peritoneal Carcinoma; Recurrent Primary Peritoneal Endometrioid Adenocarcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; olaparib; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (olaparib) (Active Comparator): Patients receive olaparib PO BID in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI as well as blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Olaparib
- Arm II (olaparib, tremelimumab) (Experimental): Patients receive olaparib as in Arm I. Patients also receive tremelimumab IV over 60 minutes on day 1. Cycles of tremelimumab repeat every 4 weeks for 4 doses and then every 12 weeks for up to 2 years total in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI as well as blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Drug: Olaparib; Biological: Tremelimumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
  Arms: Arm I (olaparib)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP 675; CP 675206; CP-675; CP-675,206; CP-675206; CP675; CP675206; Imjudo; Ticilimumab; Tremelimumab-actl
  Arms: Arm II (olaparib, tremelimumab)

SUMMARY:
This phase II trial studies how well olaparib with or without tremelimumab works in treating patients with ovarian, fallopian tube, or peritoneal cancer that has come back (recurrent). PARPs are proteins that help repair deoxyribonucleic acid (DNA) mutations. PARP inhibitors, such as olaparib, can keep PARP from working, so tumor cells can't repair themselves, and they may stop growing. Immunotherapy with monoclonal antibodies, such as tremelimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving olaparib and tremelimumab together may work better than olaparib alone in treating patients with ovarian, fallopian tube, or peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether olaparib plus tremelimumab has adequate safety in the study population. (Safety Lead-in Trial Components) II. To compare the progression-free survival (PFS) duration of olaparib monotherapy versus olaparib plus tremelimumab in women with recurrent, platinum sensitive ovarian, primary peritoneal, or fallopian tube cancer. (Phase II Trial Component)

SECONDARY OBJECTIVES:

I. To compare the overall response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 in women with recurrent, platinum sensitive ovarian, primary peritoneal or fallopian tube cancer treated with either olaparib monotherapy or olaparib plus tremelimumab.

II. To compare the overall survival (OS) of women with recurrent, platinum sensitive ovarian, primary peritoneal or fallopian tube cancer treated with either olaparib monotherapy or olaparib plus tremelimumab.

EXPLORATORY OBJECTIVES:

I. To explore whether conditions in the tumor microenvironment (as measured by gene expression signature in archived tumor samples) identify patients that benefit from combined olaparib and tremelimumab immunotherapy.

II. To explore whether mutations in BRCA1/2 genes or other evidence of homologous repair deficiency (HRD+) is prognostic and/or predictive of response to combined olaparib and tremelimumab immunotherapy.

III. To explore associations between PD1 expression in the tumor microenvironment and outcome and changes in circulating leukocyte populations.

IV. To explore the correlation between tumor mutational burden and response to olaparib and tremelimumab immunotherapy.

V. To explore the impact of olaparib and tremelimumab versus olaparib monotherapy on circulating leukocyte subsets via exploration of the immunomodulatory effects of PARP inhibition and the added impact of CTLA4 blockade in this patient population.

VI. To explore cytokine/chemokine levels using a multiplex immunoassay (Olink) and correlate these levels with clinical endpoints.

VII. To use cell-free deoxyribonucleic acid (DNA) to assess BRCA mutation status as a mechanism of acquired resistance to prior PARP inhibition and to compare with treatment efficacy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive olaparib orally (PO) twice daily (BID) in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) as well as blood sample collection throughout the trial.

ARM II: Patients receive olaparib as in Arm I. Patients also receive tremelimumab intravenously (IV) over 60 minutes on day 1. Cycles of tremelimumab repeat every 4 weeks for 4 doses and then every 12 weeks for up to 2 years total in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI as well as blood sample collection throughout the trial.

After completion of study treatment, patients are followed up monthly for 3 months, then every 3 months for 2 years, followed by every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have platinum-sensitive, recurrent high-grade serous or high-grade endometrioid (grade 3) ovarian, primary peritoneal, or fallopian tube cancer. Patients with other histologies are also eligible, provided that the patient has a known deleterious germline or somatic BRCA1 or BRCA2 mutation identified through testing at a clinical laboratory. Submission of BRCA testing results (germline and/or somatic) is required for all patients.
* Platinum-sensitive disease defined as no clinical or radiographic evidence of disease recurrence for > 6 months (or 182 days) after last receipt of platinum-based therapy. The date should be calculated from the last administered dose of platinum therapy.
* Patients must have had response (complete or partial) to their prior line of platinum therapy and cannot have had progression through prior platinum-based therapy.
* Patients must have RECIST 1.1 measurable disease. Patients with biochemical recurrence based on CA125 levels alone are not eligible.
* Prior therapy:

  * Prior chemotherapy must have included a first-line platinum-based regimen with or without consolidation chemotherapy.
  * Prior bevacizumab therapy as a component of frontline or recurrent treatment is permitted.
  * Patients may have received an unlimited number of platinum-based therapies in the recurrent setting.
  * Patients may have received up to one non-platinum-based line of therapy in the recurrent setting. Prior hormonal therapy will not be counted as this non-platinum-based line.
  * Prior treatment with a PARP inhibitor:

    * Patients may not have had a prior PARP inhibitor in the recurrent setting.
    * Prior use of a PARP inhibitor in the upfront maintenance setting is allowed for women with a confirmed BRCA1 or BRCA2 germline or somatic mutation.
    * Women who received a PARP inhibitor for maintenance therapy in the frontline setting must have received at least one other chemotherapy regimen for recurrence prior to enrolling on this trial.
    * Patients who demonstrated disease progression while on a PARP inhibitor are excluded.
  * Prior hormonal-based therapy for ovarian, primary peritoneal, or fallopian tube cancer is acceptable.
* Age >= 18.
* Body weight > 30 kg.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Absolute neutrophil count (ANC) >= 1,500/mcl (within 14 days prior to enrollment)
* Platelets >= 100,000/mcl (within 14 days prior to enrollment)
* Hemoglobin >= 10 g/dL (within 14 days prior to enrollment)

  * Note: blood transfusions are not permitted within 28 days prior to enrollment
* Creatinine =< 1.5 x institutional/laboratory upper limit of normal (ULN) (within 14 days prior to enrollment)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 14 days prior to enrollment)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 times institutional ULN (within 14 days prior to enrollment)
* Adequately controlled thyroid function, with no symptoms of thyroid dysfunction and thyroid stimulating hormone (TSH) within normal limits. Thyroid replacement therapy is permitted to achieve a TSH within normal limits.
* Patients must be able to swallow and retain oral medications and not have gastrointestinal illnesses that would preclude absorption of olaparib as judged by the treating physician.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
  * Administration of study drugs (olaparib, tremelimumab) may have an adverse effect on pregnancy and poses a risk to the human fetus, including embryo-lethality. Women of childbearing potential (WOCBP) must agree to use two (2) highly effective forms of contraception from up to 14 days prior to enrollment (for oral contraceptives), during treatment, and for 6 months after the last dose of study medication.
* Life expectancy >= 12 weeks.
* Patients with brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression. Imaging studies must have been completed no later than 14 days prior to enrollment. In addition, patients must have been successfully weaned off steroid support. Patients should not have received steroids for the treatment of brain metastases within 14 days prior to enrollment.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information.

Exclusion Criteria:

* Active infection requiring antibiotic therapy (except for uncomplicated urinary tract infections), including tuberculosis.
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; and cirrhosis. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Hormonal therapy directed at treatment for the cancer must be discontinued at least 28 days prior to enrollment. Hormone replacement therapy for symptom management is permitted.
* Any other therapy directed at treating the cancer including chemotherapy, biologic/targeted agents, and immunologic agents, unless discontinued at least 28 days prior to enrollment.
* Any radiation therapy unless discontinued at least 28 days prior to enrollment.
* Major surgical procedure within 28 days prior to enrollment.
* Current or prior use of immunosuppressive medication within 14 days before enrollment. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (i.e. intra-articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (i.e. computed tomography [CT] scan contrast allergy premedication).
* Patients with active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

  * Patients with autoimmune disease (e.g., psoriasis, extensive atopic dermatitis, severe asthma, inflammatory bowel disease [IBD], multiple sclerosis [M.S.], uveitis, vasculitis) requiring concurrent use of any systemic immunosuppressants or steroids are excluded from the study. Patients with vitiligo, mild, intermittent asthma requiring only occasional beta-agonist inhaler use, or mild localized eczema are eligible.
  * Any patient with an allogeneic (allo)-transplant of any kind is excluded, including xenograft heart valve.
  * Chronic use of immune-suppressive drugs (i.e. systemic corticosteroids) for the management of cancer or non-cancer related illnesses (i.e. chronic obstructive pulmonary disease [COPD]).
  * Note: ongoing steroid use for the management of brain metastases is not permitted.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib or tremelimumab.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the patient to give written informed consent.
* Subjects must not have evidence of bowel obstruction on imaging or symptoms consistent with a bowel obstruction. Additional workup to rule this out is not required.
* Known potent CYP3A4 inhibitors or inducers must be discontinued prior to starting treatment.
* Symptoms associated with toxicities (> Common Terminology Criteria for Adverse Event [CTCAE version (v) 5.] grade 2) caused by prior cancer therapy, excluding alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

  * Patients with grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Chair.
* Patients who are receiving any other investigational agent.
* Resting electrocardiogram (ECG) with corrected QT interval (QTc) > 470 msec on two or more time points within a 24-hour period, or a family history of long QT syndrome. If an initial ECG is within normal limits, a repeat ECG is not required.
* Patients who have previously received anti-CTLA-4 antibody therapy.
* Blood transfusions are not permitted within 28 days prior to study enrollment.
* Patients must not have signs or symptoms suggestive of myelodysplastic syndrome or acute myeloid leukemia.
* Pregnant or lactating patients
* Receipt of live attenuated vaccines within 30 days of enrollment. Note: patients, if enrolled, should not receive live vaccines while receiving study treatment and up to 30 days after the last treatment dose. Inactivated vaccines are permitted.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2026-02-21 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah F Adams, Principal Investigator — NRG Oncology
Locations (20):
- United States (20):
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Augusta University Medical Center, Augusta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - M D Anderson Cancer Center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: GY021 was opened to accrual in October of 2019. The study enrolled 61 patients from December of 2019 through March of 2021. Then the study was suspended.
Groups:
- Arm I (Olaparib): Patients receive olaparib (300 mg) PO BID in the absence of disease progression or unacceptable toxicity.
  Olaparib: Given PO
- Arm II (Olaparib, Tremelimumab): Patients receive olaparib (300 mg) twice daily until disease progression or adverse events prohibit further treatment. Patients also receive tremelimumab (750 mg)* IV over 60 minutes on day 1. Cycles of tremelimumab repeat every 4 weeks for 4 doses and then every 12 weeks for up to 2 years total in the absence of disease progression or unacceptable toxicity. *If a patient's weight falls to less than or equal to 30 kg, the patient should receive weight-based dosing equivalent to 10 mg/kg of tremelimumab every 4 weeks.
  Olaparib: Given PO Tremelimumab: Given IV
Period: Overall Study
Arm/Group | Arm I (Olaparib) | Arm II (Olaparib, Tremelimumab)
Started | 30 | 31
Completed | 23 | 16
Not Completed | 7 | 15
Not completed — Adverse Event | 4 | 9
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Still on Treatment | 2 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Arm I (Olaparib): Patients receive olaparib PO BID in the absence of disease progression or unacceptable toxicity.
  Olaparib: Given PO
- Arm II (Olaparib, Tremelimumab): Patients receive olaparib as in Arm I. Patients also receive tremelimumab IV over 60 minutes on day 1. Cycles of tremelimumab repeat every 4 weeks for 4 doses and then every 12 weeks for up to 2 years total in the absence of disease progression or unacceptable toxicity.
  Olaparib: Given PO
  Tremelimumab: Given IV
- Total: Total of all reporting groups
Arm/Group | Arm I (Olaparib) | Arm II (Olaparib, Tremelimumab) | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Customized [Count of Participants; unit: Participants]
  20 - 29 years | 0 | 0 | 0
  30 - 39 years | 0 | 0 | 0
  40 - 49 years | 2 | 1 | 3
  50 - 59 years | 4 | 4 | 8
  60 - 69 years | 12 | 18 | 30
  70 - 79 years | 9 | 6 | 15
  >= 80 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 61
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 28 | 28 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 27 | 27 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: The count of participants who have progressed or died (death due to any cause). Progression is defined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Summary of RECIST 1.1 criteria for progression for this trial: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: PFS is monitored for progression or death due to any cause, whichever occurs first. The median follow-up time is 22 months. Since the study was stopped early, the follow-up for progression-free survival was significantly reduced.
Population: All randomized patients (intent to treat)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Olaparib) | Arm II (Olaparib, Tremelimumab)
Number analyzed (Participants) | 30 | 31
Participants | 24 | 23

2. Primary Outcome: Dose-limiting Toxicity (DLT) (Safety Lead-In)
Description: The outcome measure presents the count of participants who experienced a DLT. If more than six of the first 25 patients treated with Tremelimumab and Olaparib are unable to complete at least 3 cycles of treatment due to DLTs then the study will be stopped. If not, then enrollment will continue until 45 patients are enrolled. If more than 11 of the first 45 patients treated with the combination regimen are unable to complete the first 3 cycles of treatment, then enrollment will be stopped, otherwise, the trial till proceed to the third component (i.e. a phase 2 comparison of study treatments).
Time Frame: At least 4 weeks after initiating treatment, no longer than 12 weeks (three complete treatment cycles). Maximum follow-up was 12 weeks.
Population: All patients who initiated treatment on Arm II and either 1) experienced a DLT or 2) completed three cycles. Patients randomized to Arm I are excluded from DLT assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Olaparib) | Arm II (Olaparib, Tremelimumab)
Number analyzed (Participants) | 0 | 25
Participants | 0 | 6

3. Secondary Outcome: Objective Response (RECIST 1.1)
Description: The objective response (RECIST 1.1) is the count of subjects with a best overall complete response (CR) or partial response (PR) among those with target lesions at the time of enrollment. : Summary of RECIST 1.1 criteria for progression for this trial: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: The median follow-up is 22 months. Since the study was stopped early, the follow-up time frame for objective response was significantly reduced.
Population: All randomized patients (intent to treat).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Olaparib) | Arm II (Olaparib, Tremelimumab)
Number analyzed (Participants) | 30 | 31
Participants | 11 | 9
Statistical Analysis 1: Comparison: Arm I (Olaparib) vs Arm II (Olaparib, Tremelimumab); Odds ratio for experimental arm (O + T) response compared to control arm (O) response; Test type: Superiority; Odds Ratio (OR) = 0.707, 95% CI 2-sided [0.241 to 2.068] — The numerator is the experimental arm (odds of response) and the denominator is the control arm (odds of response)

4. Secondary Outcome: Number of Participants Died
Description: Overall survival (OS) will be presented as survival events (deaths).
Time Frame: Overall survival will be monitored from enrollment to randomization to the date of death due to any cause. The median follow-up is 22 months. Since the study was stopped early, the time frame for OS follow-up was significantly reduced.
Population: All randomized patients (intent-to-treat).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Olaparib) | Arm II (Olaparib, Tremelimumab)
Number analyzed (Participants) | 30 | 31
Participants | 9 | 11

5. Secondary Outcome: Number of Participants With Adverse Event of Grade 3 or Higher
Description: Safety data will be summarized for all treated subjects. All adverse events, including severe adverse events (SAEs) and treatment-related adverse events, will be categorized and graded for severity according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. This will be presented as the count of participants who experienced an adverse event (AE) of grade 3 or higher.
Time Frame: During treatment period and up to 30 days after treatment end. The mean follow-up for adverse events was 6.4 months. Note: survival is monitored for a longer period of time (i.e. up to five years) as compared to the period for collecting adverse events.
Population: All randomized patients who initiated treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Olaparib) | Arm II (Olaparib, Tremelimumab)
Number analyzed (Participants) | 30 | 30
Participants | 15 | 20

ADVERSE EVENTS:
Time Frame: During treatment period and up to 30 days after treatment end. The mean follow-up for adverse events was 6.4 months. Note: overall survival (OS) is monitored for a longer period of time (i.e. up to five years) as compared to the period for collecting adverse events. The treatment period ends when the patient progresses or an adverse event prevents further treatments. Once the treatment period ends, adverse events will only be collected for an additional 30 days.
Description: All adverse events, including severe adverse events (SAEs) and treatment-related adverse events, will be categorized and graded for severity according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. There is one less patient in the AE/SAE section than in the All Cause Mortality section. This is due to one patient never being treated. Therefore this patient is excluded from adverse events, however this patient was still followed for survival status.
Arm/Group | Arm I (Olaparib) | Arm II (Olaparib, Tremelimumab)
All-Cause Mortality (participants affected / at risk) | 9/30 | 11/31
Serious Adverse Events (participants affected / at risk) | 15/30 | 20/30
Other Adverse Events (participants affected / at risk) | 30/30 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Olaparib) (N=30) | Arm II (Olaparib, Tremelimumab) (N=30)
Anemia (Blood and lymphatic system disorders) | 4 | 6
Sinus Bradycardia (Cardiac disorders) | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Adrenal Insufficiency (Endocrine disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 2 | 3
Peritoneal Necrosis (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 4 | 4
Edema Limbs (General disorders) | 0 | 1
Generalized Edema (General disorders) | 0 | 1
Autoimmune Disorder (Immune system disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 3
Lung Infection (Infections and infestations) | 1 | 0
Appendicitis Perforated (Infections and infestations) | 1 | 0
Gastrointestinal Anastomotic Leak (Injury, poisoning and procedural complications) | 0 | 1
Platelet Count Decreased (Investigations) | 0 | 1
Neutrophil Count Decreased (Investigations) | 2 | 0
Lymphocyte Count Decreased (Investigations) | 1 | 1
Electrocardiogram Qt Corrected Interval Prolonged (Investigations) | 1 | 0
White Blood Cell Decreased (Investigations) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Stroke (Nervous system disorders) | 2 | 2
Seizure (Nervous system disorders) | 1 | 0
Psychosis (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Thromboembolic Event (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 3 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Olaparib) (N=30) | Arm II (Olaparib, Tremelimumab) (N=30)
Anemia (Blood and lymphatic system disorders) | 19 | 17
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 3
Hypophysitis (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 4
Hypopituitarism (Endocrine disorders) | 0 | 1
Blurred Vision (Eye disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 8 | 15
Dry Mouth (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 10 | 6
Colitis (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 7 | 10
Stomach Pain (Gastrointestinal disorders) | 3 | 1
Rectal Pain (Gastrointestinal disorders) | 0 | 2
Bloating (Gastrointestinal disorders) | 1 | 4
Rectal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 15 | 21
Dysphagia (Gastrointestinal disorders) | 1 | 0
Mucositis Oral (Gastrointestinal disorders) | 4 | 3
Hemorrhoids (Gastrointestinal disorders) | 0 | 2
Fecal Incontinence (Gastrointestinal disorders) | 0 | 2
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Oral Dysesthesia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2
Abdominal Pain (Gastrointestinal disorders) | 8 | 7
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 1
Belching (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 3
Pain (General disorders) | 2 | 1
Flu Like Symptoms (General disorders) | 1 | 0
Fever (General disorders) | 0 | 3
Fatigue (General disorders) | 18 | 15
Non-Cardiac Chest Pain (General disorders) | 2 | 0
Edema Limbs (General disorders) | 2 | 1
Edema Face (General disorders) | 0 | 1
Chills (General disorders) | 2 | 2
Generalized Edema (General disorders) | 0 | 1
Autoimmune Disorder (Immune system disorders) | 1 | 0
Tooth Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 5
Thrush (Infections and infestations) | 0 | 1
Vaginal Infection (Infections and infestations) | 1 | 1
Skin Infection (Infections and infestations) | 0 | 1
Shingles (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Otitis Externa (Infections and infestations) | 0 | 1
Eye Infection (Infections and infestations) | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 2 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Burn (Injury, poisoning and procedural complications) | 0 | 1
Weight Loss (Investigations) | 5 | 3
Weight Gain (Investigations) | 1 | 1
Thyroid Stimulating Hormone Increased (Investigations) | 0 | 3
Platelet Count Decreased (Investigations) | 3 | 3
Neutrophil Count Decreased (Investigations) | 5 | 2
Lymphocyte Count Decreased (Investigations) | 2 | 3
Hemoglobin Increased (Investigations) | 0 | 1
Electrocardiogram Qt Corrected Interval Prolonged (Investigations) | 1 | 0
Creatinine Increased (Investigations) | 12 | 11
Cardiac Troponin T Increased (Investigations) | 1 | 0
Cardiac Troponin I Increased (Investigations) | 0 | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 1
Blood Bilirubin Increased (Investigations) | 0 | 2
White Blood Cell Decreased (Investigations) | 11 | 6
Aspartate Aminotransferase Increased (Investigations) | 4 | 6
Alkaline Phosphatase Increased (Investigations) | 2 | 4
Alanine Aminotransferase Increased (Investigations) | 4 | 3
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 8 | 7
Hypokalemia (Metabolism and nutrition disorders) | 5 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 5
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 3
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 6
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 3
Anorexia (Metabolism and nutrition disorders) | 9 | 9
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Stroke (Nervous system disorders) | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 3
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 0
Memory Impairment (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 7 | 11
Dysgeusia (Nervous system disorders) | 6 | 4
Dizziness (Nervous system disorders) | 2 | 5
Insomnia (Psychiatric disorders) | 3 | 3
Depression (Psychiatric disorders) | 2 | 3
Confusion (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 4 | 0
Urinary Tract Pain (Renal and urinary disorders) | 0 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1
Urinary Frequency (Renal and urinary disorders) | 4 | 3
Renal Calculi (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 1
Urinary Urgency (Renal and urinary disorders) | 0 | 2
Hematuria (Renal and urinary disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 2 | 2
Pelvic Pain (Reproductive system and breast disorders) | 2 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 3 | 7
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 6
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0
Thromboembolic Event (Vascular disorders) | 3 | 3
Hypotension (Vascular disorders) | 3 | 2
Hypertension (Vascular disorders) | 6 | 2
Flushing (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT04034927/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT04034927/ICF_001.pdf